CLINICAL TRIAL: NCT05229419
Title: Pattern of Acute Pediatric Poisoning at Assiut University Hospitals: Prospective Study
Brief Title: Pattern of Acute Pediatric Poisoning at Assiut University Hospitals
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Ahmed Abdelrahman, principal investigator, Assiut University
Other Study IDs: PAPTAUH
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2022-03

CONDITIONS: Poisoning
MeSH Terms: conditions — Poisoning | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute pediatric poisoning cases: All cases of acute pediatric poisoning of both sexes, in age group less than or equals to 18 years old will presenting to Assiut University Hospital with acute poisoning whose their adverse effects occurring following administration of single dose of a substance or multiple doses exposure within 24 hours.
  Interventions: Other: complete blood count

INTERVENTIONS:
Other: complete blood count — complete blood count will be done for corrosive cases

SUMMARY:
Acute pediatric poisoning is a common worldwide problematic emergency and represents frequent cause of emergency department admissions throughout the world. In 2017, the 35th Annual Report of the American Association of Poison Control Centers' National Poison Data System referred more than 2 million calls for cases of human exposure to toxic substance, more than 50% of them occurred in children less than 13 years old. Also, about 1030 patients less than 14 years old were acutely intoxicated and presented to the Regina Margherita Hospital in Italy from 2012 to 2017. According to Ain Shams study during the period between 2009 and 2013, acute poisoning presented to Ain Shams Poison Control Center; accounts for an estimated 38,470 case among children less than or equals to 18 years old. In the same age group mentioned above, about 760 cases admitted to Menoufia Poison Control Center during the year 2016, those between 2 and 6 years represented the highest age group.

Although pediatric poisoning represents a major and preventable cause of morbidity and mortality throughout the world, usually there is a great challenge with the management of acute pediatric poisoning due to the fact of difficult history taking, unreliable examination compared with that of an adult, in addition, pediatric patients are usually more vulnerable due to physiological difference between developmental stages. Also, the evident curiosity for the surroundings and the desire to explore and to emulate adults, make children particularly exposed to acute intoxications.

DETAILED DESCRIPTION:
In pediatric poisoning, the age, distribution, causes of poisoning and types of products involved differ between different geographical areas, even in the same area etiology and demographics of pediatric poisoning may change over the time depending on accessibility of poisoning to child, socioeconomic level, education, local beliefs, and customs. So, surveillance of epidemiology and patterns of children acute poisoning in each country is beneficial to define the scope of the problem and its management regarding prevention and treatment.

Acute pediatric poisoning may be unintentional (accidental, therapeutic error), or intentional (suicide, substance abuse). Unintentional poisoning is common in preschool age, mostly due to non-pharmaceutical agents, the most frequent agent of them is caustic ingestion according to Ain Shams Poison Control Center study. Caustic chemicals are widely distributed in our environment, caustic exposure is a lifelong and global problem associated with severe tissue and mucous membrane injuries with an estimated 80% of its exposure occurring among children. Caustic exposure is among the leading causes of mortality in those younger than 5 years, more than 15.8 cases per 100,000 children in the USA are reported annually, the situation is more severe in developing countries.

While the developed world has accurate demographic date about acute pediatric poisoning and its incidence, this major health problem is still insufficiently studied in the developing world and poorly documented. To knowledge, Assiut University Hospitals are lacking good demographic and epidemiological data regarding pediatric poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Children (under or equals to 18 years old)
* children with acute poisoning whose their adverse effects occurring following administration of single dose of a substance or multiple doses exposure within 24hours.

Exclusion Criteria:

- Any child with the following Criteria will be excluded from our study;

* Those with allergic reactions.
* Those with foreign body ingestion (coins, plastics, or toys).
* Those with chronic toxicity as lead poisoning.
* Any child with other diseases will not be involved in the study.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All cases of acute pediatric poisoning of both sexes, in age group less than or equals to 18 years old presenting to Assiut University Hospitals with acute poisoning whose their adverse effects occurring following administration of single dose of a substance or multiple doses exposure within 24 hours.
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of acute pediatric poisoning by numbers in Assiut University Hospitals. | 1/2/2022 to 31/1/2023
  All cases of acute pediatric poisoning of both sexes, in age group less than or equals to 18 years old will presenting to Assiut University Hospitals with acute poisoning whose their adverse effects occurring following administration of single dose of a substance or multiple doses exposure within 24 hours will be included.

SECONDARY OUTCOMES:
Correlation of acute poisoning in different pediatric age groups (from 0 to 18 years old) with each other as a plan for its appropriate prevention and management. | 1/2/2022 to 31/1/2023
  Determination of different causative agents by history, exposure route, if there is any time delay before coming to the hospital, clinical characteristics, whether the parent induced vomiting before seeking medical help or not, the outcome regarding mortality and morbidity, seasonal variation, and management data will be obtained. All of that data will be compared with each other in different pediatric age groups( infants < 1 year, toddlers 1-<3 years, preschool age 3-<6 years, school age 6-<12 years, adolescents 12-18 years) .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azab SM, Hirshon JM, Hayes BD, El-Setouhy M, Smith GS, Sakr ML, Tawfik H, Klein-Schwartz W. Epidemiology of acute poisoning in children presenting to the poisoning treatment center at Ain Shams University in Cairo, Egypt, 2009-2013. Clin Toxicol (Phila). 2016;54(1):20-6. doi: 10.3109/15563650.2015.1112014. PMID 26653953
- [Background] Berta GN, Di Scipio F, Bosetti FM, Mognetti B, Romano F, Carere ME, Del Giudice AC, Castagno E, Bondone C, Urbino AF. Childhood acute poisoning in the Italian North-West area: a six-year retrospective study. Ital J Pediatr. 2020 Jun 11;46(1):83. doi: 10.1186/s13052-020-00845-0. PMID 32527281
- [Background] Pianca TG, Sordi AO, Hartmann TC, von Diemen L. Identification and initial management of intoxication by alcohol and other drugs in the pediatric emergency room. J Pediatr (Rio J). 2017 Nov-Dec;93 Suppl 1:46-52. doi: 10.1016/j.jped.2017.06.015. Epub 2017 Sep 5. PMID 28886402
- [Background] Gummin DD, Mowry JB, Spyker DA, Brooks DE, Osterthaler KM, Banner W. 2017 Annual Report of the American Association of Poison Control Centers' National Poison Data System (NPDS): 35th Annual Report. Clin Toxicol (Phila). 2018 Dec;56(12):1213-1415. doi: 10.1080/15563650.2018.1533727. Epub 2018 Dec 21. PMID 30576252
- [Background] Park KS. Evaluation and management of caustic injuries from ingestion of Acid or alkaline substances. Clin Endosc. 2014 Jul;47(4):301-7. doi: 10.5946/ce.2014.47.4.301. Epub 2014 Jul 28. PMID 25133115
- [Background] Persson HE, Sjoberg GK, Haines JA, Pronczuk de Garbino J. Poisoning severity score. Grading of acute poisoning. J Toxicol Clin Toxicol. 1998;36(3):205-13. doi: 10.3109/15563659809028940. PMID 9656975
- [Background] Rafeey M, Ghojazadeh M, Sheikhi S, Vahedi L. Caustic Ingestion in Children: a Systematic Review and Meta-Analysis. J Caring Sci. 2016 Sep 1;5(3):251-265. doi: 10.15171/jcs.2016.027. eCollection 2016 Sep. PMID 27757390
- [Background] Urganci N, Usta M, Kalyoncu D, Demirel E. Corrosive substance ingestion in children. Indian J Pediatr. 2014 Jul;81(7):675-9. doi: 10.1007/s12098-013-1170-0. Epub 2013 Aug 7. PMID 23918323
- [Background] Uygun I, Aydogdu B, Okur MH, Arayici Y, Celik Y, Ozturk H, Otcu S. Clinico-epidemiological study of caustic substance ingestion accidents in children in Anatolia: the DROOL score as a new prognostic tool. Acta Chir Belg. 2012 Sep-Oct;112(5):346-54. doi: 10.1080/00015458.2012.11680850. PMID 23175922